# 5/1/2022 Texas A&M University Human Research Protection Program

### **INFORMED CONSENT DOCUMENT**

Title of Research Study: Advancing Precision Nutrition: Wearable Technology for Noninvasive **Insulin Monitoring** 

**Investigator:** Nicolaas Deutz, MD, PhD

# **Key Information:**

The following table is a concise and focused presentation of key information to assist you in understanding why you might or might not want to participate in the research. More detailed information is listed later on in this form.

| Why you are invited to take part in this study: | You are being asked to be in this study because we are recruiting young and older populations. The age range will include those healthy between 18-30 years old or 50-75 years of age. Your BMI is between 22-35 and you have the ability to walk, sit down and stand up with or without a walking assistance device. Also, you are willing to lay supine in bed for up to 9 hours and comply with the protocol. |
|---|---|
| Purpose of this study: | The purpose of this study is to develop a wearable device that can rapidly quantify the concentration of insulin and other molecular biomarkers in sweat. |
| Voluntary<br>Participation: | Your decision to be in this study is voluntary. |
| Right to<br>Withdraw from<br>Study: | If you decide to be in this study and then change your mind, you can leave the study at any time without penalty. |
| Length of<br>Study<br>Participation: | Your participation in this study will include 1 screening visit (~ 3 hours) and 1 study visit (~9 hours). |
| Study<br>Procedures: | The main procedures in the study include: Screening visit: Review the Informed Consent Form, conduct medical screening, vital signs, and body composition measurements. |
| | Study visits: Arrive fasted in the morning, the study nurse will insert an intravenous catheter in the hand that will be used for frequent blood draws. On the opposite limb, a microdialysis catheter will be placed in the forearm that will be used to administer a solution of amino acid tracers. There will also be a device which will be used to collect sweat and a microneedle patch with a microneedle applicator to the forearm. We will provide a standardized drink consisting of whey, maltodextrin and sunflower oil, flavored using vanilla sugar-free instant pudding. |



| Risks of Study<br>Participation: | The most common risks from participation in the study will be from the following procedures. Additional details are provided in the section "Are there any risks to me?" - Body composition scanning that includes X-ray - Placement of catheters may cause bruise, infection, allergic reaction, lightheadedness, nausea and possibly vomiting - Skin rash associated with an allergic reaction to microneedle, tape, or other medical disposables used for study purposes - Demographic and Socioeconomic Questions: Responding to demographic and socioeconomic questions could cause you to feel uncomfortable or upset. Please tell the study staff if you feel uncomfortable or upset while answering the questions. - Gastrointestinal problems like nausea, bloating, diarrhea, and vomiting associated with the intake of the study meal - The temperature-controlled hot box may cause minor irritation to your hand. |
|---|---|
| Benefit of<br>Study<br>Participation: | Vaso-vagal response associated with peripheral catheter placement. There is no direct benefit to you for participating, but your participation may help researchers learn more about metabolism. |
| Costs of Participation: | Aside from your time, there are no costs for taking part in the study. |
| Confidentiality of your information: | Information about you will be kept confidential to the extent permitted or required by law. |

<u>**Detailed Information:**</u> The following is more detailed information about this study in addition to the information listed above.

### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the Principal Investigator, Nicolaas Deutz, MD, PhD at 979-220-2910 or Research Staff at 979-422-1789 or email research@ctral.org.

This research has been reviewed and approved by the Texas A&M Institutional Review Board (IRB). You may talk to them at +1-979-458-4067, toll free at +1-855-795-8636, or by email at <u>irb@tamu.edu</u>., if

- You cannot reach the research team.
- Your questions, concerns, or complaints are not being answered by the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.



• You want to get information or provide input about this research.

## How many people will be in the research?

We expect about 32 people to participate in this research at our site, 16 for the younger population (ages 18 - 30 years) and 16 for the older population (ages 50 - 75 years).

## What happens if I say yes, I want to be in this research?

Your participation in this study will include 1 screening visit and 1 study visit. All visits will be scheduled at your convenience. All study procedures performed are for research purposes only and are not considered medical treatment or standard medical care. All personnel have received training for performing the research procedures but may not have a medical license. The procedures you will be asked to perform are described below.

### The screening visit

- a. This visit will last about 3 hours and takes place before the first study visit. Before any study-related tests and procedures are performed, researchers will discuss the study, its risks, benefits, and compensation with you. If you agree to participate, you will need to sign this consent form.
- b. During the screening visit, you will be asked questions about your health history and use of medication to determine eligibility.
- c. Furthermore, we will assess body weight, height, and vital signs.
- d. Body composition and bone density will be assessed by Dual energy X-ray Absorptiometry (DXA) and bioelectrical impedance analysis (BIA).
- e. Basic demographic information and daily life questionnaires will be administered.

Once the screening test results have been reviewed by the study personnel, we will contact you about participating in the study.

On the evenings before all study visits, from 10pm on, you will refrain from any food and drink intake. Drinking water is allowed. At the end of the study visits, you are allowed to eat and drink again. During the visits there will be the opportunity to watch television, and listen to music etc., as long as you remain in a lying or elevated position on the bed. We will also provide you with a meal at the end of the visit.

## The study visit:

- a. Please arrive fasted. This means no food or drink intake after 10pm the night before the visit. You will be allowed to have only water after 10pm. This visit will last approximately 9 hours.
- b. You will also receive glucose and amino acid tracers in your blood through an infusion line. This line is placed under the skin of your forearm using a microdialysis catheter (small, flexible, plastic tube). Glucose is a sugar and part of many carbohydrates. Amino acids are small parts of protein that naturally occur in food. They are labeled with stable tracers to make them a little heavier than normal so we can recognize them afterwards in the blood. <u>Stable means it is NOT radioactive</u>. Your body already has some of these tracers inside; we will



- simply elevate the amount by about 10% so that our lab machines can count them.
- c. The research nurse will place a catheter (small, flexible, plastic tube) in a vein of the arm or hand. The hand will be placed in a warmed box to increase blood flow. If the hand feels too warm, remove your hand from the box and notify study personnel. A cloth or gauze can be placed over the hand. The hand may be removed from the box between blood draws, but must be kept in the box for 10 minutes prior to the next blood draw. The total volume of blood drawn during the visit will be 4 tablespoons, or 65 ml, a total of 9 times during the study day.
- d. There will be a device with electrodes used to generate and collect sweat on your forearm. This device will be worn throughout the duration of the study day being 9 hours.
- e. Once sweat collection is started, we will also apply a microneedle patch to the forearm of the subject for 5-30 minutes duration. Microneedle patches (sensors) are small flexible sticker-like devices. They will be applied to the skin using a small spring loaded applicator to measure the chemical analytes in the dermal interstitial fluids. The microneedles will be applied to the skin and will only penetrate the top layer of skin.
- f. Before administration of the tracer solution, a baseline blood will be collected once for measurement of the natural enrichment of metabolites and neutrophil gelatinase-associated lipocalin (NGAL)/cystatin C by TAMU labs, as well as acute clinical chemistry biomarkers analyzed by Quest Diagnostics.
  - Hemoglobin A1C
  - Insulin
  - Renal function panel (Alb/BUN/Calcium/CO2/Cl/Creat/Glucose/Phosp/Potassium/Sodium/eGFR)
  - Hepatic function panel (ALT, AST, Alb, Alk Phos, Direct bili, Total Bili, Total protein)
  - Lipid panel (Total Cholesterol, HDL Cholesterol, LDL Cholesterol, Triglycerides, VLDL Cholesterol)
  - CBC (DIFF/PLT) (Hematocrit, Hemoglobin, MCV, MCH, MCHC, RBC, WBC, Platelet count, and percentage and absolute differential counts)
  - hsCRP
  - Cytokines
- g. During each visit, we will also measure your body weight.
- h. We will ask you to fill out questionnaires about your overall health and well-being.
- i. We will provide a standardized meal as a liquid drink consisting of whey, maltodextrin and sunflower oil, flavored using vanilla sugar-free instant pudding and will be asked to finish the drink in 10 minutes. This will occur 2 hours after the baseline sample collection.

All the above mentioned procedures are experimental. Results of testing are available upon your request.



# What are my responsibilities if I take part in this research?

If you take part in the research, it is important for your safety that you:

- Follow the directions of the research staff.
- Tell research staff about all medications you are taking (prescription and overthe-counter) and all of your health issues.
- Call the research staff at 979-422-1789 if you have any questions.

# What happens if I say yes, but I change my mind later?

You are free to leave the study at any time. There are no penalties and you do not lose any benefits to which you are otherwise entitled. Data that we have already collected will stay in the study database and cannot be removed in order to maintain the integrity of the research.

## Can I be removed from the research without my OK?

You may be removed from the study by the nurse or investigator when, in their opinion, any of the following situations is applicable:

- Determination that a condition developed that would interfere with the research methods, and which was not applicable at screening (e.g., illness, drugs).
- Signs and symptoms not seen at baseline or that worsen in severity during/ after intervention
- Catheters needed for research methods are removed before completion of the study day.
- You are not willing or unable to comply with the guidelines and procedures explained to you and mentioned in this Informed Consent form.

Early termination of your participation in the study, as decided by the Principal Investigator, can occur without your consent.

# What are the risks of being in this study? (Detailed Risks)

The things that you will be doing or undergoing have significant more risk than you would come across in everyday life. The discomforts and risks include the following:

- a. Glucose and amino acid tracers: The amino acid tracers are mixed under supervision of a licensed pharmacist in a certified clean room in the Human Clinical Research Building. On the study days, the tracers are filtered as they go directly into the bloodstream. The risks associated with administration include allergic reaction and infection, such as a change in body temperature, blood pressure and/or heart rate, flushing, itching, nausea, vomiting, fatigue, body ache, headache, sweating and chills. We will monitor for these side effects during the infusion and stop the study if needed.
- b. <u>Blood draws / catheterization</u>: Blood will be drawn multiple times during the long visits. You will receive saline after each blood sample is taken; you should experience no noticeable effects of the blood draws. A risk associated with having blood drawn is a low concentration of red blood cells. This might increase the need for blood transfusions. This is unlikely for you due to the low volume of blood samples needed for this study.



Furthermore, the risk of infection due to having blood drawn. This risk will be small as well, because it will be done using strict procedures to prevent infections.

In some instances, there might be a hematoma or bruise at the site of the catheters, or you might experience some pain as the vessel wall is pierced. Some individuals have a sudden drop in blood pressure in response to the placement of catheters in their arms. Symptoms may include lightheadedness, nausea, vomiting, and fainting. There are no long-term problems associated with this response. If you should have this response, you will be examined by the study nurse or physician and given the option of discontinuing the experiment. You may get a skin rash. This is associated with an allergic reaction to tape or other medical disposables used for the study. There may also be bleeding when the needles are inserted and when the catheters are removed. You will be given the option of discontinuing the experiment. If they find no reason to stop the study and you want to continue, you will be able to finish the study.

- c. <u>Use of temperature controlled box</u>: This method will be used to allow collection of blood from you, which is made "arterialized" by heating the air inside the box and around your hand to 50-55°C. In the event that you experience sensitivity to the heat, a wash cloth or gauze will be placed over the back of your hand and knuckles to avoid localized heating of the thin skin over the knuckles. Additionally, your hand may be removed from the hotbox between blood collections to improve comfort, but must be placed inside the hotbox 10 minutes prior to each blood collection.
- d. Assessment of body composition and bone mineral density by dual energy X-ray absorptiometry (DXA): This procedure is used to estimate the amount of fat mass and lean mass in your whole body and in your arms and legs and to measure bone mineral density in your spine and hip. For the DXA-scan you will be required to lie flat on a table for approximately 10 minutes while this test is being performed. The DXA-scans expose you to minimal radiation (2.5 mRem), equal to the natural atmospheric background radiation during 2 days in College Station. It is not harmful to you. All radiation doses carry a finite risk of inducing cancer or genetic disorders in a fetus. The DXA doses are such that these risks are small by comparison with the natural incidence of these conditions.
- e. <u>Demographic and Socioeconomic Questions</u>: Responding to demographic and socioeconomic questions could cause you to feel uncomfortable or upset. Please tell the study staff if you feel uncomfortable or upset while answering the questions.
- f. <u>Nutrition</u>: Gastrointestinal problems like nausea, bloating, diarrhea and vomiting associated with the intake of the study meal.
  - Although the researchers have tried to avoid risks, you may feel that some questions/procedures that are asked of you will be stressful or upsetting. You do not have to answer anything or undergo any procedures you do not want to.



## What are the costs of being in the research?

Taking part in this research study will not lead to any costs to you.

## What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study records, to people who have a need to review this information. We cannot promise complete privacy. Organizations that may inspect and copy your information include the TAMU HRPP/IRB and other representatives of this organization.

We may publish the results of this research. However, we will keep your name and other identifying information confidential.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

This would include blood specimens obtained during this study that will be stored for a minimum 7 years in laboratories, and may be used in future research upon approval of the Texas A&M University Human Research Protection Program office. These samples will be labeled with a code number and not with a name. These samples may be used to study other markers of protein metabolism and gut function. However, *no genetic* testing will occur on these samples. Please indicate whether you permit these specimens to be used in future research by selecting one of the following statements in the REDCap system:

- o I agree to allow my specimens to be stored for future research.
- o I do not agree to allow my specimens to be stored for future research.

If, in the future, you decide that you do not want the specimens used for research, please notify the Principal Investigator.

Funded/Supported By: USDA - Agricultural Research Service

## What else do I need to know?

Pictures and videos might be recorded. Photos and videos will be collected only on the skin with a magnified view, thus, it will not reveal any identity of a subject. If you become ill or get injured as a result of this study (medications, devices or procedures), you should seek medical treatment through your doctor or treatment center of choice. You should promptly tell the study doctor about any illness or injury. Texas A&M University has no program to pay for medical care for research-related injury. This does not keep you from seeking to be paid back for care required because of a bad outcome.

If you agree to take part in this research, compensation will be provided as follows:

- \$20 for screening
- \$150 for the study day



If all visits are completed, you will be compensated up to a total of \$170 for your time and effort. Compensation is provided in the form of a check. If the study must be stopped at any time, due to personal reasons or facility-related circumstances, you will be compensated for each part of the study you complete. If you choose to withdraw or are withdrawn from the study early, you will still be paid for the study visits or procedures you have already completed up to your last study day.

The financial office at Texas A&M University may be given your name, address, and Social Security Number in order to issue a check for your study participation. Study payments are considered taxable income and reportable to the IRS. A Form 1099 will be sent to you if your total payments are \$600 or more in a calendar year.

Your information and samples (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

**Signature Block for Capable Adult** 

| Your signature documents your permission to take part in this research. | |
|---|---|
| Signature of subject | Date |
| | _ |
| Printed name of subject | |
| Signature of person obtaining consent | Date |
| Printed name of person obtaining consent | |